CLINICAL TRIAL: NCT01804218
Title: Efficacy and Safety of Beta-adrenoceptor Inverse Agonist, Nadolol, in Mild Asthma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Invion, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: U01-BCM-01
Record Dates: First submitted 2013-03-01; First posted 2013-03-05 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: Mild Persistent Asthma, Uncomplicated
MeSH Terms: interventions — Nadolol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Active, nadolol (Experimental): Active
  Interventions: Drug: Nadolol

INTERVENTIONS:
Drug: Nadolol
  Arms: Active, nadolol
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to test the hypothesis that 18-22 week treatment with the inverse agonist nadolol will improve airway hyperresponsiveness in patients with mild asthma, compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

Individuals who meet all of the following criteria are eligible for enrollment as study participants:

1. Males and females with physician-diagnosed asthma between the ages of 18- 60.

2. Pre-bronchodilator FEV1 80% or greater than the predicted value

3. Baseline PC20 (based on FEV1) ≤ 4 mg/ml on methacholine challenge test.

4. Asthma Control Questionnaire Score (ACQ) <1.25

5. Baseline blood pressure ≥ 110/65mm Hg

6. Baseline pulse rate ≥ 60 beats/min.

7. Never-smoker or former-smoker < 10 pack.year and has not smoked within 1 year.

8. Able to complete diary cards and comply with study procedures.

9. Females of childbearing age may participate only if they have a negative pregnancy test, are non-lactating, and agree to practice an adequate birth control method (abstinence, combination barrier and spermicide, or hormonal) for the duration of the study.

Exclusion Criteria:

Subjects who meet ANY of the following criteria are not eligible for enrollment:

1. Inability or unwillingness of the participant to give written informed consent
2. History of upper/lower respiratory tract infection or asthma exacerbation requiring systemic steroids within 6 weeks of Visit 1
3. Use of rescue medication (e.g., albuterol) more than twice per week during the week preceding Visit 1 excluding the use of such medication as preventative prior to exercise.
4. History of hospitalization for asthma in the preceding year
5. History of intubation for asthma
6. Currently diagnosed with chronic obstructive pulmonary disease (COPD)
7. Currently taking any beta-blocker medication
8. History of adverse reaction or allergy to any beta-blocker medication
9. History of neurological, hepatic, renal, or other medical conditions that may interfere with the interpretation of data or the patient's participation in the study or may increase safety concerns
10. Current diabetes or hyperthyroidism
11. History of cardiovascular diseases including uncontrolled hypertension (BP >160/100), ischemic heart disease, congestive heart failure, valvular heart disease or cardiomyopathy
12. Known allergy or sensitivity to atropine or ipratropium bromide
13. Abnormal entry laboratory values at baseline except for the following tests, where values outside the normal limits will be acceptable as follows: Hct ≥ 30%, platelet count > 100,000, ALT and AST < 1.5 x upper normal limit
14. Known bleeding disorders, platelet count <100,000, PT or PTT > 1.5 x normal control (if participating in bronchoscopy sub-study)
15. Known allergy to lidocaine (if participating in bronchoscopy sub-study)
16. Documented or self-reported current history of alcoholism or drug abuse
17. Participation in another research trial within 30 days of starting this trial
18. Unwillingness or inability to comply with study procedures
19. Inability to swallow the study medication capsule
20. Use of any exclusion medication within the time period specified
21. Pregnant or nursing
22. Receiving allergen immunotherapy (desensitization injections)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-03; Primary Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
The change in methacholine provocative concentration causing a 20% fall (PC20) based on forced expiratory volume in 1 second (FEV1) between baseline visit and final dose dispensing visit. | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Nicola A. Hanania, MD, MS, Study Chair — Baylor College of Medicine
Locations (3):
- United States (3):
  - Washington University School of Medicine, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - Baylor College of Medicine, Houston, Texas